CLINICAL TRIAL: NCT05932797
Title: EVALUATION AND IMPLEMENTATION OF A MULTIMODAL INTERVENTION TO REDUCE SYMPTOMS OF LONG COVID/PROLONGED COVID IN THE ADULT POPULATION OF PUNTA ARENAS, CHILE.
Brief Title: Multimodal Long Covid19
Acronym: MLongCovid
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Magallanes (Other)
Collaborators: Teaching Assistance and Research Center of the University of Magallanes CADI-UMAG (Unknown); Clinical Hospital Dr. Lautaro Navarro Avaria (Unknown)
Responsible Party: Principal Investigator, Lidia M. Amarales Osorio, Principal Investigator, Universidad de Magallanes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SA22I0135
Record Dates: First submitted 2023-06-22; First posted 2023-07-06 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Long COVID-19 Syndrome
Keywords: Multimodal; Covid19
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19

STUDY DESIGN:
Intervention Model Description: Intervention model based on a clinical trial, in which the effectiveness of multimodal treatment will be evaluated in a research group through an ex ante, ex post measurement and then another follow-up measurement compared to a control group. In the first stage, focused on diagnosis, physical, neurological and mental health evaluations will be carried out, to then begin an interdisciplinary treatment process for 6 months, the second stage will be a retest evaluation using the same parameters used at the beginning, applied at the end of the intervention, and finally in the third stage, to evaluate the results with respect to a follow-up carried out 3 months after the end of the study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Active Comparator): Multimodal rehabilitation: physical, psychological and cognitive training and treatment program at the Teaching and Research Assistance Center of the University of Magellanus.
  Interventions: Other: Multimodal intervention in Long Covid19
- Control group (No Intervention): Individuals who must maintain their daily habits and/or usual care at their health center.

INTERVENTIONS:
Other: Multimodal intervention in Long Covid19 — The intervention will consist of physical, psychological, cognitive and nutritional training and treatment to be carried out at the Teaching and Research Assistance Center of the University of Magellanus (CADI UMAG), program includes 12 sessions of cognitive behavioral therapy sessions, 12 kinesic rehabilitation sessions, 12 treatment sessions per nutrition professional, 12 rehabilitation sessions with occupational therapy professional and 12 rehabilitation sessions with a speech therapist.
  Arms: Intervention group

SUMMARY:
Due to the COVID-19 pandemic, the world has seen the need to identify groups of patients who experience various effects in the medium and long term after recovering from the initial illness. These medium- and long-term effects are collectively known as the post-COVID-19 condition, Long-COVID, or prolonged COVID. Current evidence indicates, with conservative estimates, that between 10% and 20% of the population could be affected. Its nature is varied and ranges from physical conditions such as chronic fatigue, dyspnea and muscle weakness, to neurocognitive (compromised memory, decreased concentration) and psychological (anxiety, depression, anguish, stress). Early recognition and treatment of this symptom burden is essential for physical recovery and mental health. Due to its multivariate nature, it has been suggested that optimal recovery of patients' quality of life would only be achieved to the extent that their main symptoms are addressed from an interdisciplinary perspective.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria will be: Adults between 40 and 80 years of age. Individuals will be included if they have had a positive polymerase chain reaction (PCR) test diagnosis of SARS-CoV-2 virus, presence of dyspnea and/or fatigue greater than 3 months after COVID-19 diagnosis, at least 1 point higher on the modified Medical Research Council Scale (mMRC) compared to the period before infection. All participants must have no contraindications to perform the exercise and training tests and must be able to read, understand and sign the information and consent form.

Exclusion Criteria:

Individuals with one of the exclusion criteria will not be eligible for our research project these are: pulmonary embolism; absolute and relative contraindication to cardiopulmonary stress testing or physical training; severe exercise intolerance, significant cardiac arrhythmias or ischemia during low intensity exercise, severe pulmonary hypertension; severe pulmonary disease (e.g.: chronic obstructive pulmonary disease, severe COVID-19 related symptoms, severe asthma); recent cardiovascular event (cardiac decompensation, angioplasty or cardiac surgery less than 4 weeks old, valvular heart disease requiring surgical correction, pericarditis, ventricular rhythm disturbances and unstable despite treatment); renal failure requiring dialysis; Heart failure (NYHA III or IV).

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-11-18 (Estimated); Study Completion 2024-11-18 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by Cardiorespiratory Capacity | 24 months
  The primary outcome of the study will be measured by a maximal cardiopulmonary exercise test (CPET) on a cycloergometer. The protocol will be individualised and will include a 3-minute warm-up at 20 Watts, followed by an increasing workload of 10-20 W/min (depending on the participant's fitness level) until exhaustion, maintaining a cadence greater than 60 rpm. Electrocardiogram and oxygen saturation will be continuously monitored, while rating of perceived exertion and blood pressure will be measured every two minutes during the test. Continuously measured at rest, as well as during exercise and recovery: minute ventilation, oxygen consumption and carbon dioxide production. Gas exchange shall be collected on a breath-by-breath basis and expressed as a 15-second time average for analysis.

SECONDARY OUTCOMES:
Cardiorespiratory profiles | 24 months
  Fatigue Assessment Scale (FAS) - The FAS questionnaire consists of 10 questions and its objective is to investigate the presence of fatigue in a patient, its response is by means of a likert-type scale in which higher scores imply a greater degree of fatigue, its measurement parameters are based on two categories whose maximum score is 50 points. FAS scores 10 - 21: no fatigue (normal) FAS scores 22 - 50: substantial fatigue
Cardiorespiratory profiles | 24 months
  Test Time Up and GO - Its objective is to evaluate the dynamic balance, as well as the functional capacity and mobility of a person to perform activities of daily living. establishing mobility parameters in such a way that the more time used, the lower the mobility capacity. Less than 10 seconds: independent mobility. Between 10 and 20 seconds: mostly independent mobility. More than 20 seconds: reduced mobility.
Cardiorespiratory profiles | 24 months
  Six-minute walk test - The 6-minute walk test is a submaximal exercise test used to assess aerobic capacity and endurance. The distance walked for a time of 6 minutes is used as a result to compare changes in performance capacity. The more meters the patient runs, the better his cardiorespiratory functional capacity. If a patient reaches 304 meters in the 6 minutes, he achieves cardiorespiratory functional independence category, if he achieves less than that distance, a decrease in cardiorespiratory functional capacity is established.
Psychological profiles | 24 months
  Beck Anxiety Scale - consists of a 21-item self-administered instrument in which the patient is asked to report the extent to which he or she has been affected by each of the 21 symptoms described in the scale. Each item has four possible response options: not at all, mildly, moderately and severely. Values from 0 to 3 are assigned to each of the items. The values for each item are summed to obtain a total score that can range from 0 to 63 points. A total between 0 and 7 points is interpreted as a minimum level of anxiety, between 8 to 15 points corresponds to a mild level of anxiety, from 16 to 25 points is moderate anxiety and from 26 to 63 points is considered severe anxiety.
Psychological profiles | 24 months
  Beck Depression Scale - It consists of a 21-item self-administered instrument designed to assess the severity of depressive symptomatology in adults. In each of the items, the person has to choose, from a set of four alternatives ordered from least to most severe, the statement that best describes his or her state during the last two weeks, including the day on which he or she completes the instrument. As for the correction, each item is valued from 0 to 3 points depending on the alternative chosen and, after directly adding the score of each item, a total score can be obtained that varies from 0 to 63 points; thus, its categories range from minimal depression (0-13); mild depression (14-19), moderate depression (20-28) and severe depression (29-63).
Neurocognitive profiles | 24 months
  Montreal Cognitive Assessment - This instrument examines cognitive dysfunctions associated with attention, concentration, executive functions (including abstraction capacity), memory, language, visuoconstructive abilities, calculation and orientation. The maximum score is 30 points and its score is proportional to the level of cognitive functionality, so that the lower the score, the greater the cognitive impairment. A score equal to or higher than 26 points is considered normal; a score lower than 10 points implies incipient cognitive impairment; from 20 to 23 points: Mild cognitive impairment and if the patient achieves 26 points or more, there is no alteration of cognitive functions.
Functional profiles | 24 months
  Barthel Index - It is a test that provides ranges with scores between 0 and 100, regarding the level of functional behavioral independence for a patient. The closer a subject's score is to 0, the more dependent he/she is; the closer to 100, the more independent he/she is. Based on the results obtained in the evaluation with the Barthel Index or Scale, the classification will be: Total Dependent (less than 20 points), Severe Dependence (20 - 35 points), Moderate Dependence (40 - 55 points), Mild Dependence (greater than or equal to 60 points) and Independence (100 points).
Quality of life indicators | 24 months
  Short Form 12 Health Survey - Health related quality of life questionnaire. The response options of the SF-12 form Likert-type scales that evaluate intensity or frequency of quality of life indicators associated with health. The number of response options ranges from three to six, depending on the item, and each question is given a value that is then transformed into a scale from 0 to 100. The scores have a mean of 50 with a standard deviation of 10, so that values above 50 indicate better health-related quality of life or below 50 indicate a worse state of health-related quality of life.
Nutritional profile | 24 months
  Body composition analyzer - This instrument establishes the level of body fat in people, establishing frames of reference with scores differentiated by sex, classifying as low range in men when their score is less than 9.9%, and women less than 17.9%; normal level: Men between 10 to 19.9%, women between 18 to 27.9%; High: Men between 20 to 58%, women between 28.0 to 58%. Therefore, the higher the percentage, the higher the degree of health risks associated with overweight.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Magallanes, Punta Arenas, Provincia De Magallanes, Chile

IPD SHARING:
Plan to Share IPD: Yes
The data Will be Shared is all the individual participant data collected during the trial, after deidentification.
  Supporting information:
Supporting Information: Study Protocol, ICF
Time Frame: Immediately after finishing the process of treatment and follow-up, cleaning, quality control and analysis of our data, we will make them available to the research community in general. All data from data made available for public use will be de-identified data, i.e., stripped of private health information and devoid of private and protected health information that could be used to infer the identity of subjects. identity of individual subjects, in accordance with the Standard.
Access Criteria: Multimodal LongCov-19 Study website to be determined.

REFERENCES:
- [Background] Sarmiento Varon L, Gonzalez-Puelma J, Medina-Ortiz D, Aldridge J, Alvarez-Saravia D, Uribe-Paredes R, Navarrete MA. The role of machine learning in health policies during the COVID-19 pandemic and in long COVID management. Front Public Health. 2023 Apr 11;11:1140353. doi: 10.3389/fpubh.2023.1140353. eCollection 2023. PMID 37113165
- [Background] Alvarado-Aravena C, Arriaza K, Castillo-Aguilar M, Flores K, Dagnino-Subiabre A, Estrada-Goic C, Nunez-Espinosa C. Effect of Confinement on Anxiety Symptoms and Sleep Quality during the COVID-19 Pandemic. Behav Sci (Basel). 2022 Oct 17;12(10):398. doi: 10.3390/bs12100398. PMID 36285967
- [Background] Gonzalez-Puelma J, Aldridge J, Montes de Oca M, Pinto M, Uribe-Paredes R, Fernandez-Goycoolea J, Alvarez-Saravia D, Alvarez H, Encina G, Weitzel T, Munoz R, Olivera-Nappa A, Pantano S, Navarrete MA. Mutation in a SARS-CoV-2 Haplotype from Sub-Antarctic Chile Reveals New Insights into the Spike's Dynamics. Viruses. 2021 May 11;13(5):883. doi: 10.3390/v13050883. PMID 34064904